CLINICAL TRIAL: NCT03738579
Title: Assessment of the Improvement of Wound Healing Rate and Wound Bioburden With the Combination of Next Science BlastX Antimicrobial Wound Gel and TorrentX Wound Wash
Brief Title: Evaluating Wound Healing With Next Science Gel & Wash.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment
Sponsor: Next Science TM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSP-009
Record Dates: First submitted 2018-10-26; First posted 2018-11-13 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Chronic Wound
Keywords: biofilm; EPS matrix; antimicrobial
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The study model is modified psuedo-factorial design with a parallel base. The Next Science treatment arm (using TorrentX Wound Wash and BlastX Wound Gel) is compared against 2 controls, one using a standard dressing and another using a standard dressing with an antimicrobial component.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Control Group (Active Comparator): After standard of care debridement and irrigation (using normal saline), Mepilex foam dressing will be used. Foam dressing will be used throughout the study, including for mid-week dressing changes.
  Interventions: Device: Control Group
- Antibacterial Control (Active Comparator): After standard of care debridement and irrigation (using normal saline), Mepilex AG foam dressing will be used. This dressing will be used throughout the study, including for mid-week dressing changes.
  Interventions: Device: Antibacterial Control Group
- Next Science Group (Experimental): Standard of care debridement will be performed as well as irrigation using TorrentX Wound Wash,then BlastX Wound gel will be applied to the wound before covering treatment site with Mepilex foam dressing (no AG component). BlastX will re-applied again mid-week during mid-week dressing change.
  Interventions: Device: Next Science Group

INTERVENTIONS:
Device: Next Science Group — TorrentX Wound Wash will be used for irrigation and then BlastX Wound Gel will be applied to the wound after debridement/irrigation during in-clinic visits. BlastX Wound Gel will be re-applied again during mid-week dressing change. Dressing used will be plain foam dressing from control group arm.
  Other Names: TorrentX and BlastX
  Arms: Next Science Group
Device: Control Group — Foam Dressing will be used in conjunction with standard of care for chronic wound management, such as debridement and irrigation.
  Other Names: Foam Dressing; Mepilex Foam Dressing
  Arms: Control Group
Device: Antibacterial Control Group — Foam Dressing AG will be used in conjunction with standard of care for chronic wound management, such as debridement and irrigation.
  Other Names: Silver-based Foam Dressing; Mepilex Ag Foam Dressing
  Arms: Antibacterial Control

SUMMARY:
This is a 12-week, single-site, open-label prospective study in adult with a chronic wound diagnosis. Subjects will be randomized in equal numbers to either the control treatment arm, antimicrobial control treatment arm, or Next Science treatment arm and will receive this treatment until the wound is completely healed or they are exited from the study. Subjects will have a weekly in-office debridement visit for up to 12 weeks.

DETAILED DESCRIPTION:
This is a 12-week, single-site, open-label prospective study in adult subjects ages 18 years of age and older with a chronic wound diagnosis. There will be 15 completed subjects with up to 18 enrolled. Subjects will be randomized in equal numbers to control group (Mepilex Foam dressing); antimicrobial control group (Mepilex Ag Foam dressing); or Next Science group (TorrentX irrigation, BlastX application, and Mepilex foam dressing). Subjects will receive this treatment until the wound is completely healed or they are exited from the study. Subjects will have a weekly in-office debridement visit for up to 12 weeks. For the Next Science arm, TorrentX will be used during in-office debridement whereas BlastX will be applied once during the in-office visit and then mid-week with dressing change. DNA and plate count analysis will be taken at maximum of 5 time points: baseline/randomization visit, maximum of 3 treatment visits (Visits 3, 5, and 9), and Visit 13/Study exit (if applicable), with cultures taken pre- and post- debridement. Wound measurements will be taken via imaging from Silhouette camera system at every in-clinic visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years or older
2. Presence of full-thickness chronic wound for more than one month (i.e. chronic)
3. Ulcer must be greater than 1 cm2 to enable biofilm sampling
4. He/she is determined to NOT require endovascular or vascular reconstructive surgery to restore blood flow to the wound within the study period
5. Willing to comply with all study procedures and be available for the duration of the study
6. Provide signed and dated informed consent

Exclusion Criteria:

1. Subjects unable to provide signed and dated informed consent
2. Male or female less than 18 years old
3. Presence of a full-thickness chronic wound for less than one month
4. Subjects with a history of bleeding dyscrasia or with medical conditions that would make a bleeding complication likely
5. Subjects whose wound is less than 1 cm2
6. He/she requires endovascular or surgical arterial intervention during the study period
7. Subject with known allergic reaction to the study products ingredients
8. Wound, in the investigator's clinical judgment, is not amenable to management solely with the techniques described in this study (i.e., should be managed in addition with hyperbaric oxygen, vacuum suction, or other adjunctive methods)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Wound Size and Volume | 12 weeks
  Significantly Reduced Wound Size and Volume (measured using Aranz Aranz Medical Silhouette Imaging System) at One or More of the Measured Time Points with Next Science Group compared to Control Group(s)
Wound Closure | 12 weeks
  Significantly Earlier Wound Time to Closure at One or More of the Measured Time Points with Next Science Group compared to Control Group(s)

SECONDARY OUTCOMES:
Colony Forming Units | 12 weeks
  Reduction of viable bacteria in the Next Science test group at one or more of the time points compared to the control group(s) as measured by Colony Forming Units.
DNA Quantification | 12 weeks
  Reduction of bacteria in the Next Science test group at one or more of the times points compared to the control group(s) as measured by DNA quantification.
Bacterial species change | 12 weeks
  Changes in bacterial species will also be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Niezgoda, MD, Principal Investigator — Advancing the Zenith of Healthcare
Locations (1):
- Advancing the Zenith of Healthcare, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No